CLINICAL TRIAL: NCT01451632
Title: A Phase 1 Study of MM-121 in Combination With Cetuximab and Irinotecan in Patients With Advanced Cancers
Brief Title: A Safety Study of MM-121 With Cetuximab and Irinotecan in Patients With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-121-05-01-05 (TCD11696)
Record Dates: First submitted 2011-10-07; First posted 2011-10-13 (Estimated); Results first posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer; Squamous Cell Head and Neck Cancer; Non-small Cell Lung Cancer; Triple Negative Breast Cancer; Other Tumors With EGFR Dependence
Keywords: Metastatic Colorectal cancer; Kras wild-type; Squamous cell head and neck cancer; Non-small cell lung cancer; Triple negative breast cancer; EGFR; ErbB3; MM-121; Cetuximab; Irinotecan
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms | interventions — seribantumab; Irinotecan; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: MM-121 + cetuximab (Experimental): increasing doses of weekly MM-121 + weekly cetuximab
  Interventions: Drug: MM-121; Drug: Cetuximab
- Part 2: MM-121 + cetuximab + irinotecan (Experimental): increasing doses of irinotecan + the Recommended Phase 2 Dose/Maximum Tolerated Dose (RP2D/MTD) of MM121 + cetuximab as determined in Part 1
  Interventions: Drug: MM-121; Drug: Irinotecan; Drug: Cetuximab

INTERVENTIONS:
Drug: MM-121 — escalating doses MM-121 IV QW
  Other Names: Seribantumab, SAR256212
Drug: Irinotecan — 180 mg/m2 IV Q2W
  Other Names: Camptosar
  Arms: Part 2: MM-121 + cetuximab + irinotecan
Drug: Cetuximab — escalating doses cetuximab IV QW
  Other Names: Erbitux

SUMMARY:
The purpose of this study was to evaluate the safety and tolerability of escalating doses of the MM-121 plus cetuximab and the MM-121 plus cetuximab plus irinotecan combination.

DETAILED DESCRIPTION:
This study was a Phase 1 and pharmacologic dose-escalation trial of MM-121 plus cetuximab plus irinotecan. The study assessed the safety, tolerability, and pharmacokinetics of MM-121, cetuximab and irinotecan.

ELIGIBILITY:
Inclusion Criteria:

* No standard options remaining
* Adequate liver and kidney functions
* 18 years of age or above

Exclusion Criteria:

* History of any secondary active cancer in the last 3 years.
* Pregnant or breast feeding
* History of severe allergic reactions or contraindications to cetuximab or irinotecan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Moyo, MD, Study Director — Merrimack Pharmaceuticals
Locations (4):
- United States (4):
  - San Francisco, California
  - Boston, Massachusetts
  - Chapel Hill, North Carolina
  - Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Cohort 1: MM-121: 12 mg/kg IV weekly in 4-week cycles Cetuximab: 400 mg/m2 IV one-time loading dose followed by 200 mg/m2 IV weekly maintenance doses
- Part 1: Cohort 2a: MM-121: 20 mg/kg IV QW Cetuximab: 400 mg/m2 loading dose followed by 200 mg/m2 maintenance IV QW
- Part 1: Cohort 2b: MM-121: 12 mg/kg IV QW Cetuximab: 400 mg/m2 loading dose followed by 250 mg/m2 maintenance IV QW
- Part 1: Cohort 3a: MM-121: 40 mg/kg loading dose followed by 20 mg/kg IV QW Cetuximab: 400 mg/m2 loading dose followed by 200 mg/m2 maintenance IV QW
- Part 1: Cohort 3b: MM-121: 20 mg/kg IV QW Cetuximab: 400 mg/m2 loading dose followed by 250 mg/m2 maintenance IV QW
- Part 1: Cohort 4: MM-121: 40 mg/kg one time loading dose followed by 20 mg/kg IV QW Cetuximab: 400 mg/m2 one-time loading dose followed by 250 mg/m2 maintenance IV QW
- Part 1: Expansion Cohort: MM-121: 40 mg/kg loading dose followed by 20 mg/kg IV QW Cetuximab: 400 mg/m2 loading dose followed by 250 mg/m2 maintenance IV QW
- Part 2: Cohort 1: MM-121: 20 mg/kg IV QW
  Cetuximab: 400 mg/m2 loading dose followed by 200 mg/m2 maintenance IV QW
  Irinotecan: 180 mg/m2 IV Q2W
- Part 2: Cohort 2: MM-121: 40 mg/kg loading dose followed by 20 mg/kg IV QW
  Cetuximab: 400 mg/m2 loading dose followed by 250 mg/m2 maintenance IV QW
  Irinotecan: 180 mg/m2 IV Q2W
- Part 2: Expansion Cohort: MM-121: 20 mg/kg IV QW
  Cetuximab: 400 mg/m2 loading dose followed by 250 mg/m2 maintenance IV QW
  Irinotecan: 180 mg/m2 IV Q2W
Period: Overall Study
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2a | Part 1: Cohort 2b | Part 1: Cohort 3a | Part 1: Cohort 3b | Part 1: Cohort 4 | Part 1: Expansion Cohort | Part 2: Cohort 1 | Part 2: Cohort 2 | Part 2: Expansion Cohort
Started | 8 | 4 | 3 | 3 | 4 | 4 | 8 | 6 | 4 | 4
Completed | 8 | 4 | 3 | 3 | 4 | 4 | 8 | 6 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: MM-121 + Cetuximab: increasing doses of weekly MM-121 + weekly cetuximab
  MM-121 (SAR256212): MM-121 (SAR256212) (IV) plus Cetuximab (IV) and Irinotecan (IV)
  Cetuximab: MM-121 (SAR256212) (IV) plus Cetuximab (IV) and Irinotecan (IV)
- Part 2: MM-121 + Cetuximab + Irinotecan: increasing doses of irinotecan + the RP2D of MM121 + cetuximab as determined in Part 1
  MM-121 (SAR256212): MM-121 (SAR256212) (IV) plus Cetuximab (IV) and Irinotecan (IV)
  Irinotecan: MM-121 (SAR256212) (IV) plus Cetuximab (IV) and Irinotecan (IV)
  Cetuximab: MM-121 (SAR256212) (IV) plus Cetuximab (IV) and Irinotecan (IV)
- Total: Total of all reporting groups
Arm/Group | Part 1: MM-121 + Cetuximab | Part 2: MM-121 + Cetuximab + Irinotecan | Total
Number analyzed (Participants) | 34 | 14 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (14.19) | 56.6 (11.38) | 56.35 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 21 | 5 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 31 | 13 | 44
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 26 | 13 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 34 | 14 | 48

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation: To Evaluate the Safety and Tolerability of Escalating Doses of the MM-121 Plus Cetuximab and the MM-121 Plus Cetuximab Plus Irinotecan Combination
Description: To establish the safety of escalating doses of MM-121 in combination with cetuximab or in combination with cetuximab and irinotecan in order to determine the recommended phase 2 dose.. Dose-escalation conducted using standard 3+3 model to determine maximum tolerated dose. Reports of Dose-Limiting Toxicities (DLTs) were assessed to determine the MTD.
Time Frame: From date of first dose to 30 days after termination, the longest 48.1 weeks
Population: Patients participating in dose escalation
Measure: Number; unit: participants reporting DLTs
Groups:
- Part 1: Cohort 1: MM-121: 12 mg/kg IV QW Cetuximab: 400 mg/m2 loading dose followed by 200 mg/m2 maintenance IV QW
- Part 1: Cohort 4: MM-121: 40 mg/kg loading dose followed by 20 mg/kg IV QW Cetuximab: 400 mg/m2 loading dose followed by 250 mg/m2 maintenance IV QW
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2a | Part 1: Cohort 2b | Part 1: Cohort 3a | Part 1: Cohort 3b | Part 1: Cohort 4 | Part 2: Cohort 1 | Part 2: Cohort 2
Number analyzed (Participants) | 8 | 4 | 3 | 3 | 4 | 4 | 6 | 4
participants reporting DLTs | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2

2. Primary Outcome: To Further Determine the Safety Parameters of the MM-121 + Cetuximab and MM-121 + Cetuximab + Irinotecan Combination by Determining the Recommended Phase 2 Dose (RP2D) of the Combination(s) (Via Recording of Maximum Tolerated Dose (MTD)): MM-121 Doses
Description: Using a 3+3 dose escalation model, the maximum tolerated dose of each combination was determined by assessing dose-limiting toxicities in each cohort. RP2D = one dose lever lower than the MTD
  Part 1:
  Cohort 1: MM-121: 12 mg/kg MM-121 QW + Cetuximab: 400 mg/m2 loading dose/200 mg/m2 (400/200) QW maintenance Cohort 2a: MM-121: 20 mg/kg IV QW + Cetuximab: 400 / 200 mg/m2 maintenance IV QW Cohort 2b: MM-121: 12 mg/kg IV QW + Cetuximab: 400 /250 mg/m2 maintenance IV QW Cohort 3a: MM-121: 40 mg/kg loading dose followed by 20 mg/kg IV QW (40/20) + Cetuximab: 400 / 200 mg/m2 maintenance IV QW Cohort 3b: MM-121 20 mg/kg IV QW + Cetuximab: 400 /250 mg/m2 maintenance IV QW Cohort 4: MM-121: 40/20 mg/kg IV QW + Cetuximab: 400 / 250 mg/m2 maintenance IV QW
  Part 2:
  Cohort 1: MM-121: 20 mg/kg IV QW + Cetuximab: 400/200 mg/m2 maintenance IV QW + Irinotecan: 180 mg/m2 IV Q2W Cohort 2: MM-121: 40 / 20 mg/kg IV QW + Cetuximab: 400/250 mg/m2 maintenance IV QW + Irinotecan: 180 mg/m2
Time Frame: From date of first dose to 30 days after termination, the longest 48.1 weeks
Population: Number of patients participating in dose-escalation portion (excluding expansion cohort patients who were not evaluated for DLTs) MTD of cetuximab and irinotecan for the combination(s) are presented in a separate endpoint entry
Measure: Number; unit: mg/kg
Arm/Group | Part 1: MM-121 + Cetuximab | Part 2: MM-121 + Cetuximab + Irinotecan
Number analyzed (Participants) | 26 | 10
mg/kg
  MM-121 loading dose | 40 | NA — The addition of the loading dose was determined to be a maximum tolerated dose, and is not included in the RP2D
  MM-121 maintenance dose | 20 | 20

3. Primary Outcome: To Further Determine the Safety Parameters of the MM-121 + Cetuximab and MM-121 + Cetuximab + Irinotecan Combination by Determining the Recommended Phase 2 Dose (RP2D) of the Combination(s): Cetuximab and Irinotecan
Description: as for outcome 2
Time Frame: From date of first dose to 30 days after termination, the longest 48.1 weeks
Population: Number of patients participating in dose-escalation portion (excluding expansion cohort patients who were not evaluated for DLTs and thus not included in determining MTD/RP2D) NOTE: MTD of MM-121 provided in separate endpoint entry
Measure: Number; unit: mg/m2
Arm/Group | Part 1: MM-121 + Cetuximab | Part 2: MM-121 + Cetuximab + Irinotecan
Number analyzed (Participants) | 26 | 10
mg/m2
  Cetuximab loading dose | 400 | 400
  Cetuximab maintenance dose | 250 | 250
  Irinotecan | NA — Irinotecan was not administered during Part 1 | 180

4. Secondary Outcome: Objective Response Rate
Description: To determine the number of patients reporting an objective response using RECIST v 1.1 where a Partial Response (PR) is defined as >20% decrease in tumor burden from baseline and a Complete Response (CR) is defined as complete disappearance from tumor burden from baseline. Objective Response is presented as the total # patients with PR or CR.
Time Frame: Patients were assessed for objective response from time of first dose through treatment termination, the longest treatment duration being 48.1 weeks
Measure: Number; unit: participants with objective response
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2a | Part 1: Cohort 2b | Part 1: Cohort 3a | Part 1: Cohort 3b | Part 1: Cohort 4 | Part 1: Expansion Cohort | Part 2: Cohort 1 | Part 2: Cohort 2 | Part 2: Expansion Cohort
Number analyzed (Participants) | 8 | 4 | 3 | 3 | 4 | 4 | 8 | 6 | 4 | 4
participants with objective response | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

5. Secondary Outcome: Pharmacokinetics
Description: Pharmacokinetic (PK) evaluation was performed on plasma samples obtained weekly for the first six weeks of the study and then on day 1 of each additional cycle to assess pre-treatment trough concentrations of MM-121. Non-compartmental analysis (NCA) was performed to calculate standard PK parameters, including the maximum observed concentration (Cmax). Serum levels of MM-121 were measured at a central lab using an enzyme-linked immunosorbent assay (ELISA). Data is presented per dose level of MM-121 (12 mg/kg, 20 mg/kg, or 40/20 mg/kg) and per study part (Part 1 or Part 2)
Time Frame: Collections taken for all patients at Cycle 1, Week 1 at pre-infusion, at the end of the infusion, and 2.5, 4, 6 and 24 hours after starting the infusion of MM-121
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- Part 1: 12 mg/kg: MM-121 mg/kg plus cetuximab at either 400/200 mg/m2 or 400/250 mg/m2
- Part 1: 20 mg/kg: MM-121: 20 mg/kg Plus cetuximab at either 400/200 mg/m2 or 400/250 mg/m2
- Part 1: 40/20 mg/kg: MM-121: 40 mg/kg loading dose followed by 20 mg/kg weekly maintenance doses Plus cetuximab at either 400/200 mg/m2 or 400/250 mg/m2
- Part 2: 20 mg/kg: MM-121: 20 mg/kg plus cetuximab at 400/250 mg/m2 plus irinotecan at 180 mg/m2
- Part 2: 40/20 mg/kg: MM-121: 40 mg/kg loading dose followed by 20 mg/kg weekly maintenance doses plus cetuximab 400/250 mg/m2 plus irinotecan 180 mg/m2
Arm/Group | Part 1: 12 mg/kg | Part 1: 20 mg/kg | Part 1: 40/20 mg/kg | Part 2: 20 mg/kg | Part 2: 40/20 mg/kg
Number analyzed (Participants) | 11 | 8 | 15 | 10 | 4
ug/mL | 316.8 (23.6) | 611.0 (45.8) | 794.1 (58.2) | 505.8 (10.2) | 1278.2 (25)

6. Secondary Outcome: Pharmacokinetic Parameters of MM-121
Description: Pharmacokinetic (PK) evaluation was performed on plasma samples obtained weekly for the first six weeks of the study and then on day 1 of each additional cycle to assess pre-treatment trough concentrations of MM-121. Non-compartmental analysis (NCA) was performed to calculate standard PK parameters, including the AUClast. Serum levels of MM-121 were measured at a central lab using an enzyme-linked immunosorbent assay (ELISA). Data is presented per dose level of MM-121 (12 mg/kg, 20 mg/kg, or 40/20 mg/kg) and per study part (Part 1 or Part 2)
Time Frame: as for outcome 5
Population: Data presented by dose level of MM-121, regardless of the cohort (i.e. 15 patients in Part 1 were administered the 40/20 dose level of MM-121: 3 in cohort 3b, 4 in cohort 4, and 8 in the Part 1 expansion)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr* ug/mL
Arm/Group | Part 1: 12 mg/kg | Part 1: 20 mg/kg | Part 1: 40/20 mg/kg | Part 2: 20 mg/kg | Part 2: 40/20 mg/kg
Number analyzed (Participants) | 11 | 8 | 15 | 10 | 4
hr* ug/mL | 24190.5 (22.0) | 53063.1 (46.1) | 91111.9 (39.9) | 47681.5 (14.2) | 98387.7 (16.2)

7. Secondary Outcome: Immunogenicity
Description: Samples were collected to determine the presence of an immunologic reaction to MM-121 (i.e. human anti-human antibodies).
Time Frame: Samples were collected for all patients pre-dose on all cycles for duration of treatment, the longest of which was 48.1 weeks, and a collection was made post-infusion in any case of infusion reaction
Measure: Number
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2a | Part 1: Cohort 2b | Part 1: Cohort 3a | Part 1: Cohort 3b | Part 1: Cohort 4 | Part 1: Expansion Cohort | Part 2: Cohort 1 | Part 2: Cohort 2 | Part 2: Expansion Cohort
Number analyzed (Participants) | 8 | 4 | 3 | 3 | 4 | 4 | 8 | 6 | 4 | 4
Value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value

ADVERSE EVENTS:
Time Frame: AEs were collected from a patient's first dose until 30 days after treatment termination. SAEs were collected from time of informed consent until 30 days after termination. If related, events could be reported at any time after termination.
Description: All related AEs ongoing at the time of treatment discontinuation were followed until resolution. Investigators were to report any AEs/SAEs assumed to be related any time, even if occurring more than 30 days after last dose. Though different for each patient, on average, patients could be followed for related AEs/SAEs for ~1 year after termination
Arm/Group | Part 1: MM-121 + Cetuximab | Part 2: MM-121 + Cetuximab + Irinotecan
Serious Adverse Events (participants affected / at risk) | 15/34 | 6/14
Other Adverse Events (participants affected / at risk) | 34/34 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: MM-121 + Cetuximab (N=34) | Part 2: MM-121 + Cetuximab + Irinotecan (N=14)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Disease Progression (General disorders) | 1 | 0
Mucosal Inflammation (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Abdominal Abscess (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Lyphoedema (Vascular disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: MM-121 + Cetuximab (N=34) | Part 2: MM-121 + Cetuximab + Irinotecan (N=14)
Dermatitis Acneform (Skin and subcutaneous tissue disorders) | 18 | 4 — Any Relationship
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 10 | 3 — Any Relationship
Rash (Skin and subcutaneous tissue disorders) | 8 | 1 — Any Relationship
Dry Skin (Skin and subcutaneous tissue disorders) | 5 | 3 — Any Relationship
Skin Fissures (Skin and subcutaneous tissue disorders) | 5 | 1 — Any Relationship
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 4 | 4 — Any Relationship
Skin Ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 — Any Relationship
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0 — Any Relationship
Pruritis Generalized (Skin and subcutaneous tissue disorders) | 2 | 0 — Any Relationship
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 3 — Any Relationship
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 — Any Relationship
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 2 — Any Relationship
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 — Any Relationship
Nail Discoloration (Skin and subcutaneous tissue disorders) | 0 | 1 — Any Relationship
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 1 — Any Relationship
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 1 — Any Relationship
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 1 — Any Relationship
Fatigue (General disorders) | 22 | 9 — Any Relationship
Mucosal Inflammation (General disorders) | 8 | 4 — Any Relationship
Chills (General disorders) | 3 | 0 — Any Relationship
Non-Cardiac Chest Pain (General disorders) | 2 | 1 — Any Relationship
Asthenia (General disorders) | 1 | 1 — Any Relationship
Impaired healing (General disorders) | 0 | 1 — Any Relationship
Pyrexia (General disorders) | 4 | 1 — Any Relationship
Diarrhea (Gastrointestinal disorders) | 17 | 13 — Any Relationship
Stomatitis (Gastrointestinal disorders) | 9 | 5 — Any Relationship
Nausea (Gastrointestinal disorders) | 8 | 8 — Any Relationship
Abdominal Pain (Gastrointestinal disorders) | 7 | 1 — Any Relationship
Constipation (Gastrointestinal disorders) | 5 | 0 — Any Relationship
Vomiting (Gastrointestinal disorders) | 5 | 5 — Any Relationship
Dyspepsia (Gastrointestinal disorders) | 4 | 1 — Any Relationship
Dry Mouth (Gastrointestinal disorders) | 2 | 0 — Any Relationship
Hemorrhoids (Gastrointestinal disorders) | 2 | 2 — Any Relationship
Oral Pain (Gastrointestinal disorders) | 2 | 0 — Any Relationship
Cheilitis (Gastrointestinal disorders) | 1 | 1 — Any Relationship
Glossodynia (Gastrointestinal disorders) | 0 | 1 — Any Relationship
Haematochezia (Gastrointestinal disorders) | 0 | 1 — Any Relationship
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 — Any Relationship
Hypomagnesemia (Metabolism and nutrition disorders) | 18 | 5 — Any Relationship
Decreased Appetite (Metabolism and nutrition disorders) | 12 | 7 — Any Relationship
Hypokalemia (Metabolism and nutrition disorders) | 10 | 9 — Any Relationship
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 4 — Any Relationship
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 3 — Any Relationship
Dehydration (Metabolism and nutrition disorders) | 0 | 6 — Any Relationship
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3 — Any Relationship
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 — Any Relationship
Headache (Nervous system disorders) | 7 | 0 — Any Relationship
Dygeusia (Nervous system disorders) | 4 | 1 — Any Relationship
Ataxia (Nervous system disorders) | 2 | 0 — Any Relationship
Dizziness (Nervous system disorders) | 1 | 2 — Any Relationship
Peripheral Neuropathy (Nervous system disorders) | 0 | 2 — Any Relationship
Central Nervous System Lesion (Nervous system disorders) | 0 | 1 — Any Relationship
Neuralgia (Nervous system disorders) | 0 | 1 — Any Relationship
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1 — Any Relationship
Paronychia (Infections and infestations) | 9 | 0 — Any Relationship
Fungal Skin Infection (Infections and infestations) | 2 | 1 — Any Relationship
Urinary Tract Infection (Infections and infestations) | 2 | 3 — Any Relationship
Bronchitis (Infections and infestations) | 0 | 1 — Any Relationship
Nail Infection (Infections and infestations) | 0 | 1 — Any Relationship
Oral Infection (Infections and infestations) | 0 | 1 — Any Relationship
Tinea Cruris (Infections and infestations) | 0 | 1 — Any Relationship
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 | 1 — Any Relationship
Vision Blurred (Eye disorders) | 3 | 1 — Any Relationship
Conjunctivitis (Eye disorders) | 2 | 1 — Any Relationship
Lacrimation increased (Eye disorders) | 2 | 0 — Any Relationship
Ocular Hyperaemia (Eye disorders) | 1 | 1 — Any Relationship
Weight Decreased (Investigations) | 8 | 7 — Any Relationship
Blood Magnesium Decreased (Investigations) | 2 | 0 — Any Relationship
White Blood Cell Count Decreased (Investigations) | 0 | 2 — Any Relationship
Neutrophil Count Decreased (Investigations) | 0 | 1 — Any Relationship
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2 — Any Relationship
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 — Any Relationship
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 — Any Relationship
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — Any Relationship
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Any Relationship
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Any Relationship
Nasal Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Any Relationship
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — Any Relationship
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — Any Relationship
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — Any Relationship
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Any Relationship
Infusion Related Reaction (Injury, poisoning and procedural complications) | 5 | 2 — Any Relationship
Post-Procedural Swelling (Injury, poisoning and procedural complications) | 0 | 1 — Any Relationship
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 — Any Relationship
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 — Any Relationship
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 — Any Relationship
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 — Any Relationship
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 — Any Relationship
Depression (Psychiatric disorders) | 3 | 0 — Any Relationship
Insomnia (Psychiatric disorders) | 3 | 1 — Any Relationship
Anxiety (Psychiatric disorders) | 2 | 1 — Any Relationship
Confusional State (Psychiatric disorders) | 2 | 0 — Any Relationship
Pericardial effusion (Cardiac disorders) | 2 | 1 — Any Relationship
Tachycardia (Cardiac disorders) | 2 | 0 — Any Relationship
Cardiac Arrest (Cardiac disorders) | 0 | 1 — Any Relationship
Anemia (Blood and lymphatic system disorders) | 6 | 1 — Any Relationship
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 — Any Relationship
Deep Vein Thrombosis (Vascular disorders) | 2 | 0 — Any Relationship
Pollakiuria (Renal and urinary disorders) | 0 | 1 — Any Relationship

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less